CLINICAL TRIAL: NCT07105085
Title: Long-Term Outcomes of ABO-Incompatible Versus Compatible Living Donor Liver Transplantation: A Single-Center Retrospective Study
Brief Title: Long-Term Outcomes of ABO-Incompatible Versus Compatible Living Donor Liver Transplantation
Status: Terminated | Type: Observational
Why Stopped: in order to get sufficient follow-up period and judged to be gather enough subjects
Sponsor: Seoung Hoon Kim (Other Government)
Responsible Party: Sponsor-Investigator, Seoung Hoon Kim, National Cancer Center, Korea, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Other Study IDs: NCC2023-0110
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplantation; Liver Diseases
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: living donor liver transplantation — other intervention cannot be applied.

SUMMARY:
This retrospective cohort study investigates the long-term outcomes of ABO-incompatible (ABO-I) versus ABO-compatible (ABO-C) living donor liver transplantation (LDLT). A total of 511 patients at a single high-volume transplant center in Korea.

The study aims to compare overall survival and the incidence of biliary complications.

DETAILED DESCRIPTION:
This retrospective cohort study investigates the long-term outcomes of ABO-incompatible (ABO-I) versus ABO-compatible (ABO-C) living donor liver transplantation (LDLT). A total of 511 patients underwent LDLT between January 2012 and December 2022 at a single high-volume transplant center in Korea. Among them, 121 received ABO-I grafts using a rituximab-based desensitization protocol, while 390 underwent ABO-C LDLT. The study aims to compare overall survival and the incidence of biliary complications, as well as to identify risk factors specific to each group. This analysis provides insights into the long-term safety and efficacy of ABO-I LDLT in regions with low deceased donor organ availability.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who underwent LDLT at the study center from 2012 to 2022

Exclusion Criteria:

* Pediatric patients, deceased donor recipients, multi-organ transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who underwent living donor liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of biliary complications | within 10 years post-transplantation
  Statistical analyses are conducted to determine the incidence of biliary complication.

CONTACTS AND LOCATIONS:
Overall Officials: Seoung Hoon kim, MD, PhD, Principal Investigator — National Cancer Center

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are not publicly available due to institutional and ethical restrictions but are available from the corresponding author on reasonable request and with permission from the institution.

DOCUMENTS (1):
  • Study Protocol (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT07105085/Prot_000.pdf